CLINICAL TRIAL: NCT05180461
Title: A Phase-II, Randomised, Double-blind, Parallel-group Trial to Investigate Emodepside (BAY 44-4400) in Subjects With Onchocerca Volvulus Infection, Comprising: Part 1 to Investigate Safety, Tolerability, Pharmacodynamics, Pharmacokinetics and Dose-Response Relationship for Efficacy (Proof-of-Concept); Part 2 to Investigate Efficacy of Selected Doses, Safety, Tolerability and Pharmacokinetics
Brief Title: Emodepside Phase II Trial for Treatment of Onchocerciasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNDi-EMO-04; UHAS-REC A.1 [1] 20-21 (Other: UHAS Research Ethics Committee)
Record Dates: First submitted 2020-10-19; First posted 2022-01-06 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Onchocerciasis
Keywords: Helminthiasis; Filariasis; Parasitic diseases; Nematode Infections; Neglected tropical diseases; Skin Diseases, Parasitic; Skin Diseases, Infectious; River blindness; Anthelmintics; Anti-Infective Agents; Antinematodal Agents; Skin diseases; Anti-parasitic agents; Octadepsipeptide (cyclic depsipeptide)
MeSH Terms: conditions — Onchocerciasis; Helminthiasis; Filariasis; Parasitic Diseases; Nematode Infections; Neglected Diseases; Skin Diseases, Parasitic; Skin Diseases, Infectious; Onchocerciasis, Ocular; Skin Diseases | interventions — emodepside; Bay 44-4400; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking applies to Parts 1a/b and Part 2. Part 0 (Pilot Group) is Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part 0 Pilot group emodepside 15mg Once a day (OD) 1 day (Experimental): emodepside tablets 15 milligrams once a day for 1 day
  Interventions: Drug: emodepside
- Part 1 emodepside 30mg OD 1 day (Experimental): emodepside tablets 30 milligrams once a day for 1 day
  Interventions: Drug: emodepside
- Part 1 emodepside 15mg OD 7 days (Experimental): emodepside tablets 15 milligrams once a day for 7 days
  Interventions: Drug: emodepside
- Part 1 emodepside 15mg OD 14 days (Experimental): emodepside tablets 15 milligrams once a day for 14 days
  Interventions: Drug: emodepside
- Part 1 emodepside 15mg twice a day (BID) 10 days (Experimental): emodepside tablets 15 milligrams twice a day for 10 days
  Interventions: Drug: emodepside
- Part 1 placebo (Placebo Comparator): matching placebo of emodepside tablets
  Interventions: Drug: matching placebo of emodepside
- Part 2 emodepside dose regimen A (Experimental): emodepside tablets, dose regimen A selected from regimens tested in Part 1
  Interventions: Drug: emodepside; Drug: matching placebo of ivermectin
- Part 2 emodepside dose regimen B (Experimental): emodepside tablets, dose regimen B selected from regimens tested in Part 1
  Interventions: Drug: emodepside; Drug: matching placebo of ivermectin
- Part 2 ivermectin (Active Comparator): ivermectin, single oral dose of 150 micrograms per kilogram by weight
  Interventions: Drug: matching placebo of emodepside; Drug: ivermectin

INTERVENTIONS:
Drug: emodepside — emodepside tablet
  Other Names: BAY 44-4400
  Arms: Part 0 Pilot group emodepside 15mg Once a day (OD) 1 day; Part 1 emodepside 15mg OD 14 days; Part 1 emodepside 15mg OD 7 days; Part 1 emodepside 15mg twice a day (BID) 10 days; Part 1 emodepside 30mg OD 1 day; Part 2 emodepside dose regimen A; Part 2 emodepside dose regimen B
Drug: matching placebo of emodepside — emodepside matching placebo tablet
  Arms: Part 1 placebo; Part 2 ivermectin
Drug: ivermectin — ivermectin tablet (overencapsulated for blinding)
  Other Names: Mectizan; Stromectol
  Arms: Part 2 ivermectin
Drug: matching placebo of ivermectin — matching placebo of overencapsulated ivermectin tablet
  Arms: Part 2 emodepside dose regimen A; Part 2 emodepside dose regimen B

SUMMARY:
The trial evaluates safety, tolerability, pharmacodynamics, pharmacokinetics, dose-response, and efficacy of emodepside tablets, administrated as a range of dose regimens, in adults infected with Onchocerca Volvulus.

DETAILED DESCRIPTION:
There is an urgent need for a macrofilaricidal drug targeting the adult stage of Onchocerca volvulus, which could be used in individual case management and, after appropriate testing, as an alternative drug to ivermectin in Mass Drug Administration (MDA) programs.

Emodepside is a promising drug candidate to kill the adult and sexually mature Onchocerca volvulus. Emodepside was shown to be macrofilaricidal and microfilaricidal against a variety of filarial nematodes in non-clinical studies, and is a registered drug for animal health, commercialized by Bayer AG under the name of Profender® (in combination with praziquantel) or Procox® (in combination with toltrazuril).

Three Phase I trials of emodepside with single or multiple doses of emodepside have been conducted in healthy Caucasian men. The results are encouraging and support continuation of the clinical development programme of emodepside as treatment for onchocerciasis. One of these trials also enabled the selection of a field-adapted tablet formulation, suitable for use in countries endemic for onchocerciasis.

The present trial is designed in a stepwise approach starting with a proof of concept part, which is further subdivided in steps to investigate the safety, tolerability and pharmacokinetics of emodepside in the target population - Part 0 (pilot group), followed by investigations of the safety of emodepside in low and high-microfilaria carriers - Part 1a, and the dose-response relationship for efficacy of emodepside compared to placebo in microfilaria-positive patients - Part 1b. This approach allows to maximize the information regarding the safety of emodepside in the target population and to establish a dose range, in which emodepside is efficacious. Based on the information obtained from Parts 0 and 1, up to two efficacious dose regimens will be selected to carry forward into the confirmatory, active-controlled Part 2 of the trial, which will investigate the superiority of emodepside over ivermectin assessed using a clinically relevant endpoint, i.e. long-term absence of microfilariae at month 24.

ELIGIBILITY:
Inclusion Criteria for Part 1:

1. Written, signed (or thumb-printed) and dated informed consent, after having the opportunity to discuss the study with the Investigator or a delegate.
2. Men and women with Onchocerca volvulus infection, 18 to 65 years of age inclusive at time of Screening,

   1. Presence of at least 1 excisable subcutaneous nodule/onchocercoma detected on palpation
   2. O. volvulus infection diagnosed by skin snip method: documented mf-positivity on skin assessment on at least 2 out of 4 skin snips.

      * i. For Part 0: subjects with low microfilarial load, skin microfilarial density > 0 and < 10 microfilariae/mg and without ocular involvement
      * ii. For Part 1a:

        * In groups with low microfilarial load, skin microfilarial density > 0 and < 10 microfilariae/mg and without ocular involvement;
        * In groups with high microfilarial load, skin microfilarial density ≥ 10 microfilariae/mg with or without ocular involvement (only in anterior segment) or skin microfilarial density > 0 and < 10 microfilariae/mg and with ocular involvement (only in anterior segment), which must include microfilariae in the eye, i.e. onchocercal corneal opacities alone are not acceptable.
      * iii. For Part 1b:

        * positive for microfilariae
3. Body weight at Screening ≥ 40 kg
4. For women of child-bearing potential, acceptance of the requirement to use a highly effective form of birth control effective from Day 0 until at least 3 months after the final intake of IMP (Month 4 visit). Choice of birth control method must be clearly documented.

Exclusion Criteria for Part 1:

1. Participation in any studies other than purely observational studies within 3 months prior to Screening or during the study, or within 5 times the half-life of the drug in the previous clinical trial, whichever is longer (time calculated relative to final intake in previous trial) or currently in the follow-up period for any clinical trial.
2. Any vaccination within 4 weeks prior to IMP administration.
3. Acute infection and/or febrile illness requiring therapy within 14 days prior to IMP administration.
4. Administration of medication or herbal therapies as follows:

   1. Administration of any medication (with the exception of diclofenac, paracetamol, ibuprofen and aspirin) or herbal preparation within 14 days prior to IMP administration, or medicine given regularly for an existing condition;
   2. The following antifilarial therapies, or medication that may have an antifilarial effect:

      * i. ivermectin; ≤ 6 months prior to IMP administration and / or
      * ii. doxycycline; ≤ 1 year prior to IMP administration: more than 2-week course and / or
      * iii. moxidectin; ≤ 2 years prior to IMP administration.
   3. Other preventive chemotherapy, e.g. as part of an MDA programme within 14 days prior to IMP administration.
5. Presence of any clinically significant medical condition at Screening: including, but not limited to diabetes type 1 or 2; past or current history of neurological or neuropsychiatric disease or epilepsy; sickle cell disease; known human immunodeficiency virus (HIV) infection, disclosed by review of medical history or concomitant medication.
6. Presence of abnormal physical findings or laboratory values at Screening that could interfere with the objectives of the trial or the safety of the subject, in the opinion of the Investigator.
7. Clinically significant history of cardiac abnormality, and/or relevant pathological abnormalities on electrocardiography at Screening, such as atrioventricular block (PR interval above 240 msec), or prolongation of the QRS complex over 120 msec or QTc interval over 450 msec (QTcB or QTcF).
8. Blood pressure and heart rate in the supine position at Screening, outside one or more of the ranges 90-140 mmHg systolic, 60-90 mmHg diastolic; heart rate 45-100 beats/min.
9. Symptoms of orthostatic hypotension at Screening, considered clinically significant in the opinion of the Investigator.
10. History of drug or alcohol abuse.
11. Use of alcohol or drugs of abuse within 48 hours before IMP administration.
12. Abnormal laboratory results at Screening, defined as (based on the reference laboratory test ranges for the study*):

    1. White blood cell count < 3.0 x 109/L
    2. Neutrophils < 1.0 x 109 /L
    3. Lymphocytes < lower limit of normal (LLN)*
    4. Haemoglobin < 11 g/dL
    5. Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and/or alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT > 2 x upper limit of normal (ULN*) and/or bilirubin > 1.5 ULN*
    6. Fasting glucose > ULN*
    7. Potassium < LLN*
    8. Serum creatinine > ULN* and estimated Glomerular Filtration Rate (using the Modification of Diet in Renal Disease equation) < 60 mL/min
    9. Any other abnormal laboratory result corresponding to Grade 2 or above in the study grading criteria, or abnormalities considered significant in the opinion of the Investigator.
13. History of severe drug allergy, non-allergic drug reactions, severe adverse reaction to any drug, or multiple drug allergies.
14. Known hypersensitivity to any ingredient of the IMP, including the active ingredient emodepside, or to ivermectin, or to any medication used during the study (e.g. for eye examinations).
15. Blood donation within 8 weeks prior to Screening or blood transfusion received within 1 year before Screening.
16. Current hyperreactive onchodermatitis or severe manifestations due to onchocerciasis.
17. Coincidental infection with other endemic filarial parasites based on laboratory tests at Screening (Wuchereria bancrofti, Mansonella spp.).
18. Coincidental infection with Loa loa based on medical history or positive test at Screening.
19. In groups intended to include subjects without ocular involvement: ocular microfilariae or onchocercal eye lesions, assessed at Screening.
20. Ophthalmological history or conditions that could make the ocular examination difficult or represent a risk for the safety of the subject in the opinion of the Investigator, assessed at Screening, including the following (subjects will be excluded if any of the criteria are met for either eye):

    1. Ocular disease including inflammatory eye disease, uveitis, glaucoma or evidence of retinal cysticercosis;
    2. History of surgery for glaucoma and/or cataract;
    3. Evidence of corneal or conjunctival damage, with or without ocular symptoms (except corneal opacities in groups intended to include subjects with ocular involvement);
    4. Evidence of an increased risk of acute glaucoma, based on examination of anterior chamber.
    5. Evidence of ocular media opacity, including lens opacity and vitreous opacities, that make difficult ocular examination in the opinion of the Investigator;
    6. Evidence of retinal or optic nerve pathology (including age-related macular degeneration (AMD));
    7. Visual impairment of best corrected or pinhole visual acuity worse than 6/18 metres, and/or visual field defect of grade 3 (on frequency doubling technology (FDT) or worse; and/or - where ocular coherence tomography (OCT) is used - severe retinal nerve fibre layer thinning in the superior and inferior quadrant analysis on OCT of the optic nerve with a corresponding visual field defect of grade 2 (on FDT) or worse on the same eye; ; or blindness;
    8. Any microfilariae identified in the posterior segment of the eye or more than 50 microfilariae in the anterior segment.
21. Unwilling to remain within the clinical research ward for the Admission Period (for Part 0 and Part 1a), or in or nearby the clinical research ward for the in-house period (for Part 1b) or unwilling to comply with the house rules of the clinical research ward.
22. Any other past or current condition that the Investigator feels would exclude the subject from the study or that places the subject at undue risk.
23. For women of child-bearing potential (WOCBP): pregnancy (determined by date of last menstrual period and serum pregnancy test prior to first intake of IMP), or breastfeeding.
24. Unwilling or unable to comply with the requirements of the study protocol for the entire duration of the study, in the opinion of the Investigator.
25. Unable to participate in the study as per local law, if applicable.

Inclusion Criteria for Part 2:

1. Written, signed (or thumb-printed) and dated informed consent, after having the opportunity to discuss the trial with the Investigator or a delegate.
2. Men and women with Onchocerca volvulus infection, 18 to 65 years of age inclusive at time of Screening.

   1. Presence of at least 1 excisable subcutaneous nodule/onchocercoma detected on palpation.
   2. Onchocerca volvulus infection diagnosed by skin snip method: documented mf-positivity on skin assessment on at least 2 out of 4 skin snips.
3. Body weight ≥ 40 kg at Screening.
4. For women of child-bearing potential, acceptance of the requirement to use a highly effective form of birth control effective from Day 0 until at least 3 months after the final intake of IMP (Month 4 visit). Choice of birth control method must be clearly documented.

Exclusion Criteria for Part 2:

1. Participation in any studies other than purely observational studies, within 3 months prior to Screening, and during the study, or within 5 times the half-life of the drug tested in the previous clinical trial, whichever is longer (time calculated relative to last dose in the previous clinical trial) or is currently in the follow-up period for any clinical trial, or received emodepside as part of a previous clinical trial.
2. Any vaccination within 4 weeks before IMP administration.
3. Acute infection and/or febrile illness requiring therapy within 14 days prior to IMP administration.
4. Administration of medication or herbal therapies as follows.

   1. Administration of any medication (with the exception of diclofenac, paracetamol, ibuprofen and aspirin) or herbal preparation within 14 days prior to IMP administration, or medicine given regularly for an existing condition, except with the approval of the Principal Investigator;
   2. The following antifilarial therapies, or medication that may have an antifilarial effect:

   i. ivermectin; ≤ 6 months prior to IMP administration and / or ii. doxycycline; ≤ 1 year prior to IMP administration: more than 2-week course and / or iii. moxidectin; ≤ 2 years prior to IMP administration. c. Other preventive chemotherapy, e.g. as part of an MDA programme within 14 days prior to IMP administration, except with the approval of the Principal Investigator.
5. Presence of any of the following at Screening that could interfere with the objectives of the trial or the safety of the subject, in the opinion of the Investigator:

   1. Abnormal physical examination or laboratory finding;
   2. Any clinically significant medical condition. Including, but not limited to diabetes type 1 or 2, significant liver or cardiovascular disease, current or previous neurological or neuropsychiatric disease or epilepsy, active infection, sickle cell disease, known human immunodeficiency virus (HIV) infection, disclosed by review of medical history or concomitant medication.
6. Recent history of drug or alcohol abuse (within 6 months prior to IMP administration).
7. Use of alcohol or drugs of abuse within 24 hours prior to IMP administration.
8. Abnormal laboratory results at Screening, defined as (based on the reference laboratory test ranges for the study*):

   1. Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and/or alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT > 2 x upper limit of normal (ULN*) and/or bilirubin > 1.5 ULN
   2. Serum creatinine > ULN* and estimated glomerular filtration rate (using the Modification of Diet in Renal Disease equation) < 60 mL/min
9. History of severe drug allergy, non-allergic drug reactions, severe adverse reaction to any drug or multiple drug allergies.
10. Current hyperreactive onchodermatitis.
11. Known hypersensitivity to any ingredient of the IMPs, including the active ingredient emodepside, or to ivermectin, or to any medication used during the study (e.g. for eye examination).
12. Blood donation within 8 weeks prior to Screening.
13. Coincidental infection with other endemic filarial parasites based on laboratory tests at Screening (Wuchereria bancrofti, Mansonella spp.)
14. Coincidental infection with Loa loa based on medical history or positive test at Screening.
15. Ophthalmological history or conditions that could interfere with the objectives of the trial or compromise the safety of the subject in the opinion of the Investigator, assessed at Screening, including the following (subjects will be excluded if any of the criteria are met for either eye):

    1. Inflammatory eye disease, glaucoma, severe uveitis, evidence of retinal cysticercosis;
    2. History of surgery for glaucoma;
    3. Severe keratitis, and/or cataracts that interfere with visualisation of the posterior segment of the eye;
    4. Evidence of an increased risk of acute glaucoma, based on examination of anterior chamber;
    5. Evidence of ocular media opacity, including lens opacity and vitreous opacities, that make difficult ocular examination in the opinion of the Investigator;
    6. Evidence of retinal or optic nerve pathology (including age-related macular degeneration (AMD));
    7. Severe visual impairment (best corrected or pinhole visual acuity worse than 6/60 metres), severe reduction of peripheral visual fields (greater than grade 3 on frequency doubling technology (FDT)) or blindness;
    8. Any microfilariae identified in the posterior segment of the eye or more than 50 microfilariae in the anterior segment.
16. Any other past or current condition that the Investigator feels would exclude the subject from the study or place the subject at undue risk.
17. For women of child-bearing potential (WOCBP): pregnancy (based on date of last menstrual period, and pregnancy test prior to first intake of IMP) or breastfeeding.
18. Unwilling or unable to comply with the requirements of the study protocol for the entire duration of the study, in the opinion of the Investigator.
19. Unable to participate in the study as per local law, if applicable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Part 1 - absence (or presence) of live female adult worms with normal embryogenesis | 12 months
  Absence (or presence) of live female adult worms with normal embryogenesis, assessed by histological examination of nodules collected on nodulectomy
Part 1 - absence (or presence) of skin microfilariae (co-primary outcome) | 12 months
  Absence (or presence) of skin microfilariae across four skin snips
Part 2 - absence (or presence) of skin microfilariae | 24 months
  Absence (or presence) of skin microfilariae, assessed across all skin snips in a participant

SECONDARY OUTCOMES:
Part 1- absence (or presence) of live female adult worms | 12 months
  The absence (or presence) of live female adult worms, assessed by histological examination of nodules collected after nodulectomy
Part 1 - presence (or absence) of dead female adult worms | 12 months
  The presence (or absence) of dead female adult worms, assessed by histological examination of nodules collected after nodulectomy
Part 1 - Absence (or presence) of skin microfilariae | up to 12 months
  Absence (or presence) of skin microfilariae
Part 1 - reduction in skin microfilarial density | up to 12 months
  The reduction in skin microfilarial density, defined as the mean number of microfilariae per milligram per subject, at all time-points after treatment related to baseline: change and percentage reduction
Part 1 - Absence (or presence) of microfilariae in nodular tissue | 12 months
  The absence (or presence) of microfilariae in nodular tissue assessed by histological examination of nodules collected after nodulectomy
Part 2 - Absence (or presence) of live female adult worms with normal embryogenesis | 24 months
  Absence (or presence) of live female adult worms with normal embryogenesis assessed by histological examination of nodules collected after nodulectomy.
Part 2 - Absence (or presence) of live female adult worms | 24 months
  Absence (or presence) of live female adult worms, assessed by histological examination of nodules collected after nodulectomy
Part 2 - Presence (or absence) of dead female adult worms | 24 months
  Presence (or absence) of dead female adult worms, assessed by histological examination of nodules collected after nodulectomy
Part 2 - Absence (or presence) of skin microfilariae | up to 24 months
  Absence (or presence) of skin microfilariae
Part 2 - The reduction in skin microfilarial density | up to 24 months
  The reduction in skin microfilarial density, defined as the mean number of microfilariae per milligram per subject, at all time-points after treatment related to baseline: change and percentage reduction
Part 2 - Absence (or presence) of microfilariae in nodular tissue | 24 months
  The absence (or presence) of microfilariae in nodular tissue, assessed by histological examination of nodules collected on nodulectomy

CONTACTS AND LOCATIONS:
Locations (3):
- Democratic Republic of the Congo (2):
  - Centre de santé de référence de Kimpese, Kimpese, Bas-Congo Province
  - Hôpital général de référence de Masimanimba, Masi-Manimba, Kwilu
- University of Health and Allied Services School of Public Health, Hohoe, Volta Region, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Summary results will be shared once Clinical Study Report will be available
Supporting Information: Study Protocol
Time Frame: Within 12 months of Clinical Study report finalization
Access Criteria: Open Access